CLINICAL TRIAL: NCT00517504
Title: Methylphenidate Study in Young Children With Developmental Disorders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC03-59
Record Dates: First submitted 2007-08-15; First posted 2007-08-17 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-07

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: methylphenidate; ritalin; attention deficit hyperactivity disorder; developmental disorder; preschool children
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Developmental Disabilities | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Methylphenidate — * 1-week single blind placebo lead-in phase.
  * step-wise single blind titration of MPH at 1.25 mg bid for the first week, 2.5 mg bid for the second week , 5 mg bid for the third week, 7.5 mg bid for the fourth week and 10 mg bid for the 5th week.
  Dose increased if room for improvement in child's symptoms and no clinically important side effects. Dose not increased if no room for improvement in child's symptoms or if clinically important side effects.
  After single blind titration, child enters a 4-week double-blind randomized crossover study with placebo and child's best dose that produced maximal effect with minimal side effects, with each child serving as his/her own control.

SUMMARY:
The purpose of this study is to determine if methylphenidate (a common brand name is Ritalin), a medicine used for treating older children with Attention Deficit and Hyperactivity Disorder (ADHD), is also safe and helpful for problems related to symptoms of ADHD in young children with Developmental Disorders (DD)

DETAILED DESCRIPTION:
Currently, there is no systematic empirical information to guide the use of methylphenidate (a common brand name is Ritalin) to treat symptoms of ADHD in young children with Autistic Disorder/Asperger's Disorder/Pervasive Developmental Disorder, Not Otherwise Specified/Developmental Disorders. Preliminary data from a recent study of ADHD in young children suggest that methylphenidate may be useful in children with developmental disorders (DD). The purpose of this study is to determine the safety and efficacy of methylphenidate to treat ADHD symptoms in young children with Pervasive Developmental Disorders (PDD) or Developmental Disorders (DD).

All subjects will be screened for eligibility inclusion and exclusion criteria. All concurrent non-pharmacological therapies will be stabilized for a minimum period of 2 weeks prior to the child's entry into the drug phase of the study. At each medication follow-up visit, a detailed history will be obtained and recorded for all concurrent treatments. If a child enrolls in this study, his/her participation will last approximately 3 to 4½ months with 12-18 outpatient daytime visits.

Screening assessment: The child's parent and teacher/daycare provider, if applicable, will need to complete some forms that describe the child's problems with overactivity, impulsivity and inattention. If these forms indicate that the child may have ADHD the investigator will schedule outpatient-screening assessments. The research staff will evaluate the child to see if s/he has a Developmental Disorder (DD) or PDD and ADHD. Each child will receive a developmental assessment, and each parent will be interviewed about his or her child's behavior. The child's teacher will be given several rating forms to complete. The parents will be asked to complete some questions about the child's development. Both parents (if available) will be interviewed about their family histories. Some of the screening assessments will be videotaped/audiotaped. Each child will have a physical examination, an electrocardiogram (EKG), a urine test and a blood test. The doctor will ask the parents about his or her child's medical history.

Medication phase: After screening assessments are completed, the child will enter the medication phase of the study. Each child will first have a step-wise single-blind titration of MPH to determine his/her best dose followed by a double-blind crossover trial with placebo and the child's best dose. The order of active drug and placebo will be randomized across the sample so that half the children will first receive MPH for 2 weeks and the other half will first receive placebo for 2 weeks. The children will receive the alternative drug condition (placebo or the child's best dose) for the next 2 weeks.

The child and his/her parents will come back each week for a clinic visit. At each visit the child's height, weight, blood pressure and pulse will be checked. The child's parents and teacher/daycare provider, if applicable, will be asked to complete some rating scales every week.

ELIGIBILITY:
Inclusion Criteria:

* 36-84 month old children
* Child must meet the DSM-IV criteria for AD or PDD NOS as determined via a parent interview on the ADI-R and on child observation via the ADOS, or DD.
* Child must have categorical and dimensional evidence of clinically significant ADHD symptoms in multiple settings that have been present for at least six months

Exclusion Criteria:

* Child with prior failed treatment with an adequate trial of methylphenidate;
* Concurrent treatment with other medications that have CNS effects or that affect performance (e.g., antidepressants, antipsychotics, alpha-agonists, adrenergic blockers, lithium carbonate, sedating antihistamines, decongestant or sympathomimetics);
* Child with a current history of chronic tic disorder (e.g., Tourette syndrome with current severity of moderate or more), or a family history of Tourette's Disorder. Children with chronic mild tics will be eligible for the study;
* Child who has a major medical condition that would interfere with involvement in the study or would be affected negatively by methylphenidate (i.e., heart disease, high blood pressure, glaucoma, untreated or unstable hyperthyroidism, uncontrolled seizure disorder, or illnesses that would require hospitalization). Children with seizures will be eligible for the study if the seizure medication is stable for 3 months and the child is seizure-free for at least 6 months;
* Child with co-morbid psychiatric diagnoses of Major Depression, Bipolar Disorder, a psychotic disorder, Rett's Disorder, Childhood Disintegrative Disorder, or other psychiatric disorders in addition to PDD and ADHD that may require treatment with additional/alternative medication;
* Current history of physical, sexual, or emotional abuse;
* The patient has taken an investigational drug within the last 30 days.

Ages: 36 Months to 84 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2001-05; Primary Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
- Hyperactive-Impulsive subscale of the Conners Rating Scale-Revised completed at baseline and at each week of the drug trial. - Clinician's Global Improvement completed at baseline and at each week of the drug trial. | 3 to 4.5 months

SECONDARY OUTCOMES:
-Hyperactive subscale of the Nisonger-Child Behavior Rating Form. -Children's Global Assessment Scale -Weekly side effect ratings and safety measures -Behavioral observation -Neuropsychological executive functions -Childhood Autism Rating Scale | 3 to 4.5 months

CONTACTS AND LOCATIONS:
Overall Officials: Jaswinder K Ghuman, M.D., Principal Investigator — University of Arizona